CLINICAL TRIAL: NCT03710382
Title: The WE Pilot Study: Walking Epidurals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 18.213
Record Dates: First submitted 2018-10-12; First posted 2018-10-18 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-01

CONDITIONS: Labor Pain
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Intervention Model Description: Prospective pilot study with single group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Walking epidural (Experimental): Parturients will receive a lower concentration of bupivacaine in their epidural infusion and will be encouraged to walk during labor.
  Interventions: Other: Walking epidural

INTERVENTIONS:
Other: Walking epidural — Parturients in spontaneous or induced labor will receive combined spinal-epidural analgesia (CSE) using an infusion of bupivacaine 0.0625% and fentanyl 2 mcg/mL and will be encouraged to walk a minimum of 15 minutes every hour during the first stage of labor.

SUMMARY:
The primary objective of the study is to assess the feasibility of a walking epidural protocol in our center. This study will provide a small data set for a larger prospective randomized controlled study.

Hypothesis: Walking a minimum of 15 minutes per hour will decrease the incidence of instrumental deliveries (forceps and vacuum) in women presenting in spontaneous or induced labor with neuraxial analgesia. Before testing this hypothesis in a randomized controlled study, the feasibility of this protocol needs to be assessed since allowing laboring women to ambulate while receiving neuraxial analgesia is not the standard-of-care at our institution.

DETAILED DESCRIPTION:
Historically, women have labored in the upright position and it is only in the twentieth century that hospitalization and bedrest have become the standard of care during labor in most developed countries. This practice has been especially encouraged in patients laboring under neuraxial analgesia (epidural or combined spinal-epidural) because of the possibility of lower limb weakness associated with the use of local anesthetic agent.

Walking during labor has been associated with positive outcomes such as a reduction in the duration of labor, reduced incidence of assisted vaginal delivery and reduction of the rate of caesarean section in women in upright position compared to those bedridden, without being associated with negative effects on mothers' and babies' well-being. Proposed hypothesis to explain the reduction in duration of labor are an improved uterine contractility and an enhancement of pelvic diameter.

Impacts of ambulation during labor have also been studied in women with neuraxial analgesia but unfortunately, in these studies, a significant proportion of patients allowed to walk did not and, if they did, the time spent ambulating was extremely variable.

The reluctance to allow women to walk during neuraxial analgesia is mainly because of concerns of a possible motor block and of orthostatic hypotension. The combination of a low dose of local anesthetic agent and of an opioid for CSE has been shown to provide good analgesia while minimizing impairment of lower limbs' strength. Since a certain degree of leg weakness can occur even with low concentrations of local anesthetic agent, it is recommended to evaluate the presence of a motor block before allowing ambulation with neuraxial analgesia. For safe ambulation, meeting the following conditions is generally recommended: no lower limb weakness, ability to perform straight leg raise and complete hip flexion, performance of a partial knee bend, ability to step up on a stool with both legs, trial of walking witnessed by a member of the staff.

The other major concern related to ambulatory neuraxial analgesia is the risk of fall secondary to hypotension. Hypotension mainly occurs at initiation of neuraxial analgesia and is usually easily treated with small doses of phenylephrine and ephedrine, giving additional intravenous fluids and by placing the patient in the full lateral position. Interestingly, blood pressure seems to be more stable in the ambulant parturient than in the supine one probably due to the reduced incidence of aortocaval compression when standing. Since hypotension is mainly seen after initiation of neuraxial analgesia, most studies will allow at least 30 minutes after the bolus injection of the local anesthetic agent and blood pressure is verified in the erect position before ambulation is allowed.

In the absence of obstetrical contraindications, walking during labor with neuraxial analgesia is safe if a low concentration of local anesthetic agents is used and in the absence of motor block and orthostatic hypotension. In addition to these conditions, women ambulating must be accompanied by a companion at all times.

Considering the benefits of the upright position during labor in women without neuraxial analgesia, investigators presume that providing neuraxial analgesia that preserves motor function and allows the parturient to walk may be of benefit regarding the duration of labor, mode of delivery and maternal satisfaction. To this day, no study with a strict protocol for walking has addressed the effect of ambulation on obstetrical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age of 37 weeks or more
* Spontaneous ou induced labor
* Singleton fetus in the vertex presentation
* Agreement from obstetrician

Exclusion Criteria:

* American Society of Anesthesiologists' classification of 3 or more
* Contraindication to epidural anesthesia
* Complicated or high-risk pregnancy or delivery
* Comorbidities preventing safe ambulation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2019-03-22 (Actual); Study Completion 2019-03-22 (Actual)

PRIMARY OUTCOMES:
Adherence of the participants to an established time of ambulation during the first stage of labor (at least 15 minutes per hour) | From the installation of the epidural catheter until complete cervical dilation, on Day 1
  Patients will be encouraged to be mobile at least 15 minutes per hour during the first stage of labor. Time spent walking or on the exercise ball will be calculated every hour.

SECONDARY OUTCOMES:
Safety of walking epidurals defined as the absence of motor block and orthostatic hypotension | Every hour, from the installation of the epidural catheter until complete cervical dilation, on Day 1
  Motor block will be assessed using the Modified Bromage Scale which is a 6-point scale where 1 means complete block (unable to move feet of knees) and 6 means able to perform partial knee bend. Hypotension will be defined as a 20% reduction in systolic blood pressure from Baseline (installation of the epidural catheter).
Quality of pain relief using a verbal numeric pain scale | Every hour, from the installation of the epidural catheter until delivery, on Day 1
  A verbal numeric pain (VNPS) scale will be used every hour to assess pain relief during the first stage of labor. On this scale, 0 means no pain and 10 means the most intense pain imaginable.
Satisfaction of the labor ward nurses towards the walking epidural protocol | Following delivery, on Day 1
  Nurses will be asked to grade their satisfaction towards the walking epidural protocol using a satisfaction scale. This is a 0 to 10 scale, where 0 means completely dissatisfied and 10 means completely satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Louise Roy, MD, FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided